CLINICAL TRIAL: NCT01517412
Title: A 24-week, Open-label, Randomized, 2-arm Parallel Group, Multinational, Multi-center Clinical Trial to Compare the Efficacy and Safety of Lixisenatide Injected Prior to the Main Meal of the Day Versus Lixisenatide Injected Prior to Breakfast in Type 2 Diabetic Patients Not Adequately Controlled on Metformin
Brief Title: Comparison of Lixisenatide Injected Prior to the Main Meal of the Day Versus Prior to Breakfast in Type 2 Diabetic Patients on Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12261; 2011-002416-85 (EudraCT Number); U1111-1118-0841 (Other: UTN)
Record Dates: First submitted 2012-01-16; First posted 2012-01-25 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Metformin; Drug Administration Routes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide Main Meal (Experimental): Lixisenatide 10 mcg once daily (QD) within 1 hour before "main meal of the day" for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 24.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Self-injector pen device (OptiClik®); Drug: Metformin
- Lixisenatide Breakfast (Active Comparator): Lixisenatide 10 mcg QD within 1 hour before "breakfast" for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 24.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Self-injector pen device (OptiClik®); Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: Solution for injection; Route of administration: Subcutaneous
Device: Self-injector pen device (OptiClik®)
Drug: Metformin — To be kept at stable dose (≥1.5 g/day) throughout the study.
  Other Names: Route of administration: Oral

SUMMARY:
Primary Objective:

- To compare the two treatment regimens in terms of change of glycosylated hemoglobin (HbA1c) from baseline to endpoint (Week 24)

Secondary Objective:

* To assess the effect of the 2 lixisenatide regimens on:

  * The percentage of participants who reached the target of HbA1c < 7% or ≤ 6.5% at Week 24
  * Fasting Plasma Glucose (FPG)
  * 7-point Self-Monitored Plasma Glucose (SMPG) profiles
  * Body weight
* To assess the safety and tolerability of the 2 lixisenatide regimens

DETAILED DESCRIPTION:
The maximum study duration was 28 weeks per participant, including a 24-week randomized treatment period.

ELIGIBILITY:
Inclusion criteria:

* Participants with type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit
* Metformin treatment at a stable dose of at least 1.5 g/day for at least 3 months prior to screening visit.

Exclusion criteria:

* Screening HbA1c < 7.0% and > 10.0%
* Fasting plasma glucose at screening > 250 mg/dL (> 13.9 mmol/L)
* Treatment with glucose-lowering agent(s) other than metformin in a period of 3 months prior to screening, previous use of insulin
* Participants who usually did not eat breakfast
* Type 1 diabetes mellitus
* Body Mass Index (BMI) ≤ 20 kg/m^2 and > 40 kg/m^2
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method
* Amylase and/or lipase > 3 times the upper limit of the normal laboratory range ( ULN) at screening
* Alanine aminotransferase (ALT) > 3 ULN at screening
* Calcitonin ≧ 20 pg/ml (5.9 pmol/L) at screening
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predisposes to MTC (e.g. multiple endocrine neoplasia syndromes)
* Any contra-indication related to metformin
* Any previous treatment with lixisenatide

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (82):
- United States (17):
  - Investigational Site Number 840112, Glendale, Arizona
  - Investigational Site Number 840113, Mesa, Arizona
  - Investigational Site Number 840105, Phoenix, Arizona
  - Investigational Site Number 840102, Tempe, Arizona
  - Investigational Site Number 840107, Tempe, Arizona
  - Investigational Site Number 840116, Mission Viejo, California
  - Investigational Site Number 840103, Northridge, California
  - Investigational Site Number 840118, Redlands, California
  - Investigational Site Number 840104, Temecula, California
  - Investigational Site Number 840122, Chicago, Illinois
  - Investigational Site Number 840119, Chicago, Illinois
  - Investigational Site Number 840114, Springfield, Illinois
  - Investigational Site Number 840120, Flint, Michigan
  - Investigational Site Number 840115, Billings, Montana
  - Investigational Site Number 840101, Sea Girt, New Jersey
  - Investigational Site Number 840111, Fargo, North Dakota
  - Investigational Site Number 840110, West Jordan, Utah
- Canada (11):
  - Investigational Site Number 124102, Brampton
  - Investigational Site Number 124108, Coquitlam
  - Investigational Site Number 124106, Etobicoke
  - Investigational Site Number 124113, Kelowna
  - Investigational Site Number 124110, Laval
  - Investigational Site Number 124103, Newmarket
  - Investigational Site Number 124101, Oakville
  - Investigational Site Number 124111, Saint Romuald
  - Investigational Site Number 124104, Thornhill
  - Investigational Site Number 124105, Toronto
  - Investigational Site Number 124112, Vancouver
- Czechia (6):
  - Investigational Site Number 203104, Pilsen
  - Investigational Site Number 203102, Prague
  - Investigational Site Number 203101, Prague
  - Investigational Site Number 203105, Prague
  - Investigational Site Number 203103, Trutnov
  - Investigational Site Number 203106, Újezd u Brna
- France (4):
  - Investigational Site Number 250108, Clermont-Ferrand
  - Investigational Site Number 250102, Menton
  - Investigational Site Number 250103, Nanterre
  - Investigational Site Number 250105, Rennes
- Germany (7):
  - Investigational Site Number 276103, Aßlar
  - Investigational Site Number 276102, Bad Mergentheim
  - Investigational Site Number 276107, Berlin
  - Investigational Site Number 276101, Heidelberg
  - Investigational Site Number 276104, Künzing
  - Investigational Site Number 276105, Pirna
  - Investigational Site Number 276108, Saint Ingbert-Oberwürzbach
- Poland (8):
  - Investigational Site Number 616106, Bytom
  - Investigational Site Number 616102, Gdansk
  - Investigational Site Number 616101, Krakow
  - Investigational Site Number 616103, Lublin
  - Investigational Site Number 616108, Oświęcim
  - Investigational Site Number 616105, Wroclaw
  - Investigational Site Number 616104, Wroclaw
  - Investigational Site Number 616107, Wroclaw
- Romania (5):
  - Investigational Site Number 642101, Bucharest
  - Investigational Site Number 642105, Oradea
  - Investigational Site Number 642102, Ploieşti
  - Investigational Site Number 642104, Reşiţa
  - Investigational Site Number 642103, Timișoara
- Russia (9):
  - Investigational Site Number 643103, Moscow
  - Investigational Site Number 643101, Moscow
  - Investigational Site Number 643106, Nizhny Novgorod
  - Investigational Site Number 643107, Saint Petersburg
  - Investigational Site Number 643105, Saint Petersburg
  - Investigational Site Number 643110, Saint Petersburg
  - Investigational Site Number 643102, Samara
  - Investigational Site Number 643108, Vladimir
  - Investigational Site Number 643104, Voronezh
- Spain (8):
  - Investigational Site Number 724107, A Coruña
  - Investigational Site Number 724104, Barcelona
  - Investigational Site Number 724103, Barcelona
  - Investigational Site Number 724102, Ferrol
  - Investigational Site Number 724101, Hostalets de Balenyà
  - Investigational Site Number 724106, Málaga
  - Investigational Site Number 724108, Segovia
  - Investigational Site Number 724105, Seville
- Ukraine (7):
  - Investigational Site Number 804108, Kharkiv
  - Investigational Site Number 804105, Kharkiv
  - Investigational Site Number 804102, Kiev
  - Investigational Site Number 804103, Kyiv
  - Investigational Site Number 804104, Mykolaiv
  - Investigational Site Number 804106, Poltava
  - Investigational Site Number 804101, Zaporozhie

REFERENCES:
- [Result] Ahren B, Vorokhobina N, Souhami E, Demil N, Ye J, Aronson R. Equal improvement in glycaemia with lixisenatide given before breakfast or the main meal of the day. J Diabetes Complications. 2014 Sep-Oct;28(5):735-41. doi: 10.1016/j.jdiacomp.2014.05.012. Epub 2014 Jun 5. PMID 25012990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 82 centers in 10 countries. A total of 734 participants were screened between February 15, 2012 and October 16, 2012. 283 participants were screen failures; main reason for screen failure was that glycosylated hemoglobin (HbA1c) values were out of protocol defined range. 451 participants were randomized.
Pre-assignment Details: Participants were stratified according to main meal of day (breakfast, lunch or dinner) and screening values of HbA1c (<8% or ≥8%).
Groups:
- Lixisenatide Main Meal: Lixisenatide 10 mcg subcutaneous (SC) injection once daily (QD) within 1 hour before "main meal of the day" for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 24 on top of metformin.
- Lixisenatide Breakfast: Lixisenatide 10 mcg SC injection QD within 1 hour before "breakfast" for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 24 on top of metformin.
Period: Overall Study
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Started | 225 | 226
Completed | 189 | 202
Not Completed | 36 | 24
Not completed — Adverse Event | 10 | 11
Not completed — Lack of Efficacy | 10 | 5
Not completed — Poor compliance to protocol | 8 | 3
Not completed — Other than specified above | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Lixisenatide Main Meal: Lixisenatide 10 mcg SC injection QD within 1 hour before "main meal of the day" for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 24 on top of metformin.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast | Total
Number analyzed (Participants) | 225 | 226 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.6) | 57.5 (9.7) | 56.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 129 | 253
  Male | 101 | 97 | 198
Race [Number; unit: participants]
  Caucasian/White | 211 | 211 | 422
  Black | 4 | 8 | 12
  Asian/Oriental | 10 | 7 | 17
Ethnicity [Number; unit: participants]
  Hispanic | 11 | 12 | 23
  Non-Hispanic | 214 | 214 | 428
Number of Participants with Categorical Body Mass Index (BMI) [Number; unit: participants]
  <30 kg/m^2 | 51 | 60 | 111
  ≥30 kg/m^2 | 174 | 166 | 340
BMI, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 33.47 (4.50) | 32.77 (4.62) | 33.12 (4.57)
HbA1c [Mean (Standard Deviation); unit: Percentage of hemoglobin] | 7.85 (0.76) | 7.93 (0.78) | 7.89 (0.77)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — N=225, 225
  mmol/L | 9.22 (2.03) | 9.31 (2.04) | 9.26 (2.03)
Average 7-point Self-monitored Plasma Glucose (SMPG) [Mean (Standard Deviation); unit: mmol/L] — N=211, 207
  mmol/L | 9.41 (2.01) | 9.71 (2.13) | 9.56 (2.07)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.69 (4.92) | 7.78 (5.56) | 7.24 (5.27)
Metformin Daily Dose [Mean (Standard Deviation); unit: mg] | 2040.7 (390.0) | 2091.2 (1255.3) | 2066.0 (929.6)
Randomization Strata of Main Meal of the Day [Number; unit: participants]
  Breakfast | 20 | 20 | 40
  Lunch | 116 | 117 | 233
  Dinner | 89 | 89 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: Change in HbA1C was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using last observation carried forward (LOCF). On-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. Here, number of participants analyzed = participants with baseline and at least one post-baseline HbA1c assessment during on-treatment period.
Time Frame: Baseline, Week 24
Population: Modified intent-to-treat (mITT) population: all randomized participants who received at least one dose of study drug and had both baseline and at least one post-baseline assessment of any primary or secondary efficacy endpoints, irrespective of compliance with study protocol and procedures.
Measure: Least Squares Mean (Standard Error); unit: Percentage of hemoglobin
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 218 | 222
Percentage of hemoglobin | -0.65 (0.074) | -0.74 (0.074)
Statistical Analysis 1: Comparison: Lixisenatide Main Meal vs Lixisenatide Breakfast; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of screening HbA1c (<8.0%, ≥8.0%), randomization strata of main meal of the day and country as fixed effects and baseline HbA1c value as a covariate; Test type: Non-Inferiority or Equivalence — A step-down procedure was used to control the type I error: non-inferiority of lixisenatide prior to the main meal of the day versus lixisenatide prior to breakfast was tested first. If non-inferiority was established, then a test of superiority of lixisenatide prior to the main meal of the day over lixisenatide prior to breakfast was to be performed. The non-inferiority was assessed using upper bound of 2-sided 95% CI at a level of ≤0.4%; Least square (LS) mean difference = 0.09, 95% CI 2-sided [-0.067 to 0.242], Standard Error of Mean 0.079 — Lixisenatide Main Meal vs Lixisenatide Breakfast
Statistical Analysis 2: Comparison: Lixisenatide Main Meal vs Lixisenatide Breakfast; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of screening HbA1c (<8.0%, ≥8.0%), randomization strata of main meal of the day and country as fixed effects and baseline HbA1c value as a covariate. A step-down procedure was used to control the type I error. The superiority was assessed by comparing the p-value at significance level = 0.05; Test type: Superiority or Other; p = 0.2664, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = 0.09, Standard Error of Mean 0.079 — Lixisenatide Main Meal vs Lixisenatide Breakfast

2. Secondary Outcome: Percentage of Participants With HbA1c Level <7 % or ≤6.5% at Week 24
Description: Here, number of participants analyzed = participants with baseline and at least one post-baseline HbA1c assessment during on-treatment period.
Time Frame: Week 24
Population: mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 218 | 222
Percentage of participants
  HbA1c <7% | 43.6 | 42.8
  HbA1c ≤6.5% | 22.5 | 25.7

3. Secondary Outcome: Change in Average 7-point SMPG Profiles From Baseline to Week 24
Description: Participants recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime two times in a week before baseline, before visit Week 8, before visit Week 12 and before visit week 24. The average value across the profiles performed in the week a visit for the 7-time points was calculated. Change in average 7-point SMPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to the day of last dose of study drug. Here, number of participants analyzed = participants with baseline and at least one post-baseline 7-point SMPG assessment during on-treatment period.
Time Frame: Baseline, Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 202 | 200
mmol/L | -0.80 (0.145) | -1.10 (0.145)

4. Secondary Outcome: Change in FPG From Baseline to Week 24
Description: Change in FPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to 1 day after the last dose of study drug. Here, number of participants analyzed = participants with baseline and at least one post-baseline FPG assessment during on-treatment period.
Time Frame: Baseline, Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 220 | 222
mmol/L | -0.35 (0.192) | -0.57 (0.193)

5. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 3 days after the last dose of study drug. Here, number of participants analyzed = participants with baseline and at least one post-baseline body weight assessment during on-treatment period.
Time Frame: Baseline, Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 220 | 224
kg | -2.60 (0.320) | -2.80 (0.319)

6. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7% at Week 24 And Did Not Experience Confirmed Symptomatic Hypoglycemia (Plasma Glucose [PG] <60 mg/dL [3.3 mmol/L]) During 24-Week Treatment Period
Description: Symptomatic hypoglycemia was defined as an event with clinical symptoms that were considered to result from hypoglycemic episode with an accompanying PG<60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate if no PG measurement was available. On-treatment period for symptomatic hypoglycemia assessment was defined as time from first dose of study drug up to 1 day after last dose of study drug. Participants without any post-baseline on-treatment value for HbA1c were counted as non-responders if they experienced at least one symptomatic hypoglycemia. Otherwise, they were counted as missing.
Time Frame: Week 24
Population: mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 218 | 222
Percentage of participants | 40.4 | 41.0

7. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7% And Had No Body Weight Gain at Week 24
Description: Participants without post-baseline on-treatment values for (HbA1c and body weight) that were no more than 30 days apart were counted as non-responders if at least one of the components (HbA1c and/or body weight) was available and showed no response. Otherwise, they were counted as missing.
Time Frame: Week 24
Population: mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 218 | 223
Percentage of participants | 40.8 | 38.6

8. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7% And Had No Body Weight Gain at Week 24 And Did Not Experience Confirmed Symptomatic Hypoglycemia (PG<60 mg/dL [3.3 mmol/L]) During the 24-Week Treatment Period
Description: Participants without post-baseline on-treatment values (for HbA1c and body weight) that were no more than 30 days apart not more than 30-days apart were counted as non-responders if at least one of components (HbA1c and/or body weight) was available and showed no response. Otherwise, they were counted as missing.
Time Frame: Week 24
Population: mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 218 | 223
Percentage of participants | 38.1 | 37.2

9. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7% And Had a 2-hour Postprandial Plasma Glucose (PPG) <140mg/dL After Breakfast or Main Meal At Week 24
Description: On-treatment period for 2-hour PPG assessment was defined as the time from the first dose of study drug up to the day of last dose of study drug. Participants without post-baseline on-treatment values (for HbA1c and 2-hour PPG) that were no more than 30-days apart were counted as non-responders if at least one of the components (HbA1cand/or 2-hour PPG) was available and showed no response. Otherwise, they were counted as missing.
Time Frame: Week 24
Population: mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 218 | 221
Percentage of participants | 28.9 | 27.6

10. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire Score (DTSQs) From Baseline to Week 24
Description: DTSQ is a validated measure to assess how satisfied participants with diabetes are with their treatment and how they perceive hyper- and hypoglycemia. It consists of 8 questions which are answered on a Likert scale from 0 to 6. DTSQ treatment satisfaction score is the sum of question 1, 4, 5, 6, 7 and 8 scores and ranges between 0 and 36, where higher scores indicate more treatment satisfaction. On-treatment period for treatment satisfaction assessment was defined as the time from the first dose of study drug up to 3 days after the last dose of study drug. Missing data was imputed using LOCF. Here, number of participants analyzed = participants with both baseline and Week 24 DTSQ score assessment during on-treatment period.
Time Frame: Baseline, Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Number analyzed (Participants) | 204 | 215
Units on a scale | 3.01 (0.546) | 3.54 (0.529)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 171) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported adverse events are treatment-emergent adverse events that developed/worsened during the 'on treatment period' (time from the first dose of study drug up to 3 days after the last dose of study drug). Safety population defined as all randomized participants who received at least one dose of study drug.
Arm/Group | Lixisenatide Main Meal | Lixisenatide Breakfast
Serious Adverse Events (participants affected / at risk) | 7/225 | 7/226
Other Adverse Events (participants affected / at risk) | 65/225 | 60/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide Main Meal (N=225) | Lixisenatide Breakfast (N=226)
Cellulitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide Main Meal (N=225) | Lixisenatide Breakfast (N=226)
Nasopharyngitis (Infections and infestations) | 22 | 16
Hypoglycaemia (Metabolism and nutrition disorders) | 15 | 7
Headache (Nervous system disorders) | 8 | 16
Nausea (Gastrointestinal disorders) | 33 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.